CLINICAL TRIAL: NCT04448288
Title: Time-based Effects of Stretching on Hamstrings Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal investigator, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RRC-2019-003
Record Dates: First submitted 2020-05-06; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Stretch
Keywords: Stretching; Muscle strength; Hamstring Muscles
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hamstring Group (Experimental): Pretest-posttest experimental design. Subjects participated in three experimental trials on three different days. On day-I for static-stretching for 2 minutes (SS2), day-II for 4 minutes (SS4), and day-III for 8 minutes (SS8). Testing was conducted before (pre), immediately after (post), and at 10 and 20 min post stretching. MVCF was measured using strain gauze as main outcome measure. The SS trials involved varied repetitions of 30-s static-stretches and 20-s relax period. MVC force was assessed.
  Interventions: Other: Static stretching

INTERVENTIONS:
Other: Static stretching — Static stretchings were performed by subjects that involved varied repetitions of 30-s static-stretches and 20-s relax period.

SUMMARY:
Stretching is reported to have detrimental effects on strength and thus avoided prior to strength training session. Do stretching indeed decreases muscle strength? To examine the time course (immediate, 10- and 20-min post stretching) for the effects of 2, 4, and 8 min long duration of static-stretching (SS) on isometric maximum voluntary contraction (MVC) force of hamstring muscles.

DETAILED DESCRIPTION:
OBJECTIVE: To examine the time course (immediate, 10- and 20-min post stretching) for the effects of 2, 4, and 8 min long duration of static-stretching (SS) on isometric maximum voluntary contraction (MVC) force of hamstring muscles.

METHODS: Pretest-posttest experimental design. Total of 14 subjects with mean age 25 years participated in three experimental trials on three different days. On day-I for static-stretching for 2 minutes (SS2), day-II for 4 minutes (SS4), and day-III for 8 minutes (SS8). Testing was conducted before (pre), immediately after (post), and at 10 and 20 min post stretching. MVCF was measured using strain gauze as the main outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects used to engage in 1 to 5 hours of physical activity per week. They were not doing stretching exercises regularly.

Exclusion Criteria:

* Subjects having any current injury specific to lower limb joints or current neuromuscular disease were excluded from the study.

Ages: 24 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Change in Maximum voluntary contraction force (MVCF) before and after stretching | MVCF was measured on 3 different days with each day separated by 3-4 days.
  Change in Isometric strength (MVCF) was measured before and after stretching using strain gauge

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, MPTh, Principal Investigator — Rehabilitation research chair
Locations (1):
- King Saud University, Riyadh, Saudi Arabia